CLINICAL TRIAL: NCT04852263
Title: Using a Shortened Uncuffed Endotracheal Tube as a Nasopharyngeal Airway: a Useful Adjunct During Fiberoptic Intubation Training Among Anesthesia Residents
Brief Title: Shortened Uncuffed Endotracheal Tube as a Nasopharyngeal Airway in Training in Fiberoptic Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Ahmed Abodonya, Assistant Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC-HSD-67-2021
Record Dates: First submitted 2021-04-09; First posted 2021-04-21 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Other): Fiberoptic intubation was carried out without nasopharyngeal airway
  Interventions: Other: Group I
- Group II (NPA group) (Other): Fiberoptic intubation was performed with a modified nasopharyngeal airway.
  Interventions: Other: Group II (NPA group)

INTERVENTIONS:
Other: Group I — Oral fiberoptic intubation was carried out using lingual traction without nasopharyngeal airway.
  Other Names: Oral fiberoptic intubation
  Arms: Group I
Other: Group II (NPA group) — Oral fiberoptic intubation was carried out using lingual traction plus modified nasopharyngeal airway.
  Other Names: Oral fiberoptic intubation plus modified nasopharyngeal airway
  Arms: Group II (NPA group)

SUMMARY:
Background: Fiberoptic intubation is an effective technique for establishing airway access in patients with critical airways.

Objective: It was hypothesized that the learning of oral fiberoptic intubation by the anesthesia resident trainee is easier and safe using modified nasopharyngeal airway.

Methodology: This prospective randomized study was done on 62 adult patients with normal airway scheduled for elective oral fiberoptic intubation, their age 20 -60 years, 56 males and 6 females, American Society of Anesthesiologists I-III class. After institute ethical committee clearance and written informed consent, patients were randomly divided into two groups of 31 each; Group I: oral fiberoptic intubation was carried out using lingual traction. In group II, FOI was carried out using lingual traction plus a shortened uncuffed nasal endotracheal tube (modified nasopharyngeal airway). Time taken to successful tracheal intubation and other technical parameters were recorded. Heart rate, mean arterial blood pressure, oxygen saturation, end-tidal carbon dioxide tension, and any associated complications were also recorded.

DETAILED DESCRIPTION:
Patients with normal airway, 20 - 60 years, ASA grade I-III with mallampati class I or II were scheduled for elective oral FOI. Patients who refused to undergo the procedure, presence of an absolute contraindication to nasal intubation like head trauma, a nasal mass, and deviated nasal septum were excluded from the study.

Patients were randomly divided into two equal groups; Group I: FOI was carried out without NPA, and Group II: FOI was performed using NPA (NPA group). Lingual traction was used in both groups. Patients were optimized for surgery and fasting for 8 hours. While the patients in the preoperative holding area, they were premedicated with glycopyrrolate 0.2 mg intravenously 30 min prior to the procedure. At the same time, patients have been treated with xylometazoline 0.1% nasal drops in both nostrils followed by lignocaine jelly 2%.

All staff in the pre, intra, and postoperative area are licensed with ACLS according to the standard and guidelines of patient safety. The patient file and vital signs will be monitored during the stay in the holding area to discover any abnormalities. And each patient will sign a written consent form after explaining and informing about the procedure of the study. Vital signs (pulse, blood pressure, respiratory rate, and body temperature) and oxygen saturation will be checked before receiving any medication and frequently every 5 minutes till the end of the procedure to detect early concerns (hemodynamics instability, bleeding, neurocognitive dysfunction, and failed technique) The procedure was stopped if any patient feels abnormality or observed by a physician.

ENT consultant must be informed before the procedure to be around. Consultant Anesthesia will be closely included during the procedure for maintaining the accurate and optimum procedure.

In the operating room, patients were connected to standard monitors including pulse oximetry, ECG, non-invasive blood pressure, and temperature monitoring prior to administering premedication drugs. Then, 2 mg of midazolam and 50 μg fentanyl were injected intravenously 3 min prior to the procedure. In a group, II (NPA group), when the patient sedated with midazolam and fentanyl, a well-lubricated uncuffed tube (Portex®) 7.0 for male and 6.5 for female) was inserted nasally and advanced until the tip stands just above the opening of the larynx and then connected to a source of oxygen. After a period of 2-3 min of preoxygenation, the patient was anesthetized with total intravenous anesthesia (TIVA) using propofol and remifentanil infusion. The anesthesia resident trainee was asked to use a fiberoptic bronchoscope (Karl Storz® Intubation fiberscope 11301 BN1) to pass it through a cuffed endotracheal tube (ETT), visualize the vocal cords, pass through the glottic aperture and then pass the ETT over the fiberoptic bronchoscope. The correct ETT placement was confirmed by visualization of the carina and tracheal rings and bilateral equal air entry. The same scenario was done by the resident trainee in group I but without using the NPA.

The time of fiberscope insertion and intubation and the number of attempts were recorded. Hemodynamic and respiratory changes (HR, MAP, SpO2, and ETCo2) were recorded at 3 points; at the baseline before induction of anesthesia, during insertion of the scope (two minutes after induction of anesthesia), and after FOI (two minutes after securing ETT). Any adverse events were also recorded as sore throat, PONV, dental trauma,...etc. If necessary, facilitating techniques like jaw thrusts were used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal airway,
* 20-60 years,
* ASA grade I - III with mallampati class I or II.

Exclusion Criteria:

* Patients who refused to undergo the procedure,
* Presence of an absolute contraindication to nasal intubation like head trauma, a nasal mass, and deviated nasal septum.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | During procedure
  It was regularly observed during procedure

SECONDARY OUTCOMES:
Time taken to successful intubation | During procedure
  It was recorded from starting to completion of fibroptic intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sattam bin Abdulaziz University, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided